CLINICAL TRIAL: NCT06679036
Title: An Open, Multicenter Phase Ib/II Clinical Study on the Safety, Tolerance, Pharmacokinetics, and Initial Efficacy of HRS-2189 in Combination With Fluvastatin±HRS-6209, or HRS-8080±HRS-6209, or HRS-6209+HRS-1358 in Patients With Advanced Unresectable or Metastatic Breast Cancer
Brief Title: A Trial of HRS-2189 in Combination With Fluvastatin±HRS-6209, or HRS-8080±HRS-6209, or HRS-6209+HRS-1358 in Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-2189-201-BC
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Advanced Unresectable or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group A (Experimental): HRS-2189 in combination with Fluvustat.
  Interventions: Drug: HRS-2189; Drug: Fluvustat
- Treatment group B (Experimental): HRS-2189 in combination with HRS-8080.
  Interventions: Drug: HRS-2189; Drug: HRS-8080
- Treatment group C (Experimental): HRS-2189 in combination with HRS-6209 and Fluvustat.
  Interventions: Drug: HRS-2189; Drug: Fluvustat; Drug: HRS-6209
- Treatment group D (Experimental): HRS-2189 in combination with HRS-6209 and HRS-8080.
  Interventions: Drug: HRS-2189; Drug: HRS-8080; Drug: HRS-6209
- Treatment group E (Experimental): HRS-2189 in combination with HRS-6209 and HRS-1358.
  Interventions: Drug: HRS-2189; Drug: HRS-6209; Drug: HRS-1358

INTERVENTIONS:
Drug: HRS-2189 — HRS-2189
Drug: Fluvustat — Fluvustat
  Arms: Treatment group A; Treatment group C
Drug: HRS-8080 — HRS-8080
  Arms: Treatment group B; Treatment group D
Drug: HRS-6209 — HRS-6209
  Arms: Treatment group C; Treatment group D; Treatment group E
Drug: HRS-1358 — HRS-1358
  Arms: Treatment group E

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of dexmedetomidine hydrochloride nasal spray for preoperative sedation in adults. To explore the reasonable dosage of dexmedetomidine hydrochloride nasal spray for preoperative sedation.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG physical condition 0-1 point.
2. Advanced unresectable or metastatic breast cancer confirmed by histopathology or cytopathology.
3. Menopausal Status.
4. Previous treatments: (New) adjuvant endocrine therapy combined or not combined with CDK4/6 inhibitors during or within 12 months after treatment, including recurrence/metastasis, shall be counted as one line of endocrine therapy and one line of CDK4/6 inhibitor therapy (such as combined CDK4/6 inhibitors); Relapse/metastasis during (new) adjuvant chemotherapy or within 6 months after the end of treatment (whichever occurs later), counted as one line of chemotherapy.
5. Disease progression confirmed by imaging during or after the last systemic anti-tumor treatment before the first use of medication (limited to the stage of efficacy expansion).
6. There must be at least one measurable extracranial lesion that meets RECIST v1.1 at baseline.
7. Expected survival>3 months.
8. The functional level of 8 organs is good.
9. Previous treatments: The interval between receiving nitrosourea or mitomycin C before the first medication in this study was ≥ 6 weeks; Receiving cytotoxic drugs, endocrine therapy, immunotherapy, targeted therapy, surgical interval (excluding biopsy or PICC catheterization or PORT infusion port catheterization surgery), or other clinical studies with the last dose of medication ≥ 4 weeks; The interval between the end of radiotherapy is ≥ 2 weeks.
10. female participants with fertility must agree to use efficient contraceptive measures for contraception during the study treatment period and within 7 months after the end of the study treatment period; Female subjects with fertility must have a negative serum HCG test within 7 days prior to enrollment in the study and must be non lactating.
11. Voluntarily participate in this clinical trial, willing and able to comply with the clinical visit and research related procedures, understand the research procedures, and have signed informed consent.

Exclusion Criteria:

1. Patients with active (uncontrolled or symptomatic) brain metastases, cancerous meningitis, spinal cord compression, or a history of primary CNS tumors; patients with brain metastases who have completed treatment at least 28 days prior to first use of the study drug and are asymptomatic can be considered for enrollment if they have been confirmed asymptomatic by cranial imaging studies such as CT, MRI, or venography without evidence of cerebral hemorrhage, and have completed treatment at least 28 days before the first use of the study drug.
2. Patients with a history of severe cardiovascular disease, including: (1) Congestive heart failure (NYHA Class>2); (2) Severe/unstable angina, new angina within the last 3 months; (3) Myocardial ischemia requiring long-term medication control; patients with NYHA Class III-IV heart failure; (4) Acute myocardial infarction within the last 6 months; (5) Any grade 2 or higher supraventricular or ventricular arrhythmia that requires treatment or intervention; (6) Atrial fibrillation, coronary/peripheral artery bypass grafts, or cerebrovascular symptoms including transient ischemic attacks.
3. Patients with factors affecting oral medication intake, such as difficulty swallowing or intestinal obstruction, or have active gastrointestinal diseases or other diseases that may significantly affect drug absorption, distribution, metabolism, or excretion (active inflammatory bowel disease or chronic diarrhea, enterocolitis or upper gastrointestinal surgery, including gastrectomy).
4. Patients with uncontrollable third space effusions (such as large ascites, pleural effusion, pericardial effusion) or cancerous lymphedema.
5. Pregnant women, nursing mothers, or those planning to become pregnant during the study period.
6. Patients with significant liver disease history, untreated active hepatitis B (defined as positivity for HBsAg or HBcAb and HBV-DNA levels above the normal upper limit), or active hepatitis C (defined as HCV-RNA levels above the detection limit).
7. Patients with uncontrolled chronic systemic comorbidities (such as severe chronic lung, liver, kidney or heart diseases).
8. Patients with active autoimmune diseases, history of immune deficiency, autoimmune disease history, or history of diseases or syndromes requiring systemic corticosteroid hormones or immunosuppressive drug therapy, or have acquired (HIV infection) or congenital immunodeficiency diseases, or have a history of organ transplantation (including homologous bone marrow transplantation).
9. Patients with active infectious tuberculosis and need for antimicrobial treatment.
10. Patients with known significant liver disease history, untreated active hepatitis B (defined as positivity for HBsAg or HBcAb and HBV-DNA levels above the normal upper limit), or active hepatitis C (defined as HCV-RNA levels above the detection limit).
11. Patients who have had other malignancies within the past 5 years, except: 1) Completely cured skin basal cell carcinoma and cervical intraepithelial neoplasia; 2) Completely cured and without recurrence of secondary primary cancer within 5 years.
12. Patients who have used strong or moderate inhibitors of CYP3A4 within 1 week before the first dose or strong or moderate inducers of CYP3A4 within 2 weeks before the first dose.
13. Pregnant women, nursing mothers, or those planning to become pregnant during the study period.
14. Patients with a history of neurological or psychiatric disorders, or those with a history of abuse of psychotropic drugs or drug addiction.
15. Patients who are expected to receive other anti-tumor treatments or medications during this study.
16. Patients with other serious physical or laboratory abnormalities that may increase the risk of participating in the study or interfere with study results, and those deemed by the investigator not suitable for participation in this study.
17. Patients with anti-tumor treatment-related toxicity in the past (excluding alopecia; according to the judgment of the investigator， after consultation with the sponsor, some tolerable chronic Grade II toxicities may be excluded).
18. Patients who have an allergy to any study drug or any excipient.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs+SAEs | From the first drug administration to within 30 days for the last treatment dose.
Dose limited toxicity (DLT) | Up to 28 days.
Maximum tolerated dose (MTD) | Up to 28 days.
Recommended Phase II Dose (RP2D) | Up to 28 days.
ORR (objective response rate) - Stage II (efficacy expansion) | Every 8 weeks lasting about one year.

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter: Cmax,ss | 2 months.
Evaluation of pharmacokinetic parameter: Tmax,ss | 2 months.
Evaluation of pharmacokinetic parameter: Cmin,ss | 2 months.
Evaluation of pharmacokinetic parameter: AUCss | 2 months.
Best Overall Response (BOR) | Every 8 weeks lasting about one year.
Duration of Response (DoR) | Every 8 weeks lasting about one year.
Disease Control Rate (DCR) | Every 8 weeks lasting about one year.
Clinical Benefit Rate (CBR) | Every 8 weeks lasting about one year.
Progression Free Survival (PFS) | Every 8 weeks lasting about one year.
Changes in antibody levels in PBMCs relative to baseline | 1 month.
Evaluate the correlation between target amplification and clinical efficacy | From the first drug administration to within 30 days for the last treatment dose.
Evaluation of the correlation between gene mutations in ctDNA and clinical efficacy, as well as the mechanism of drug resistance. | From the first drug administration to within 30 days for the last treatment dose.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Harbin Medical University Affiliated Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided